CLINICAL TRIAL: NCT05835921
Title: Enhancing Prospective Thinking in Early Recovery
Acronym: RENTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Brandon G. Oberlin, PhD, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1805574553; Aims 5-6; RENTS (Other: IndianaU); 1R34DA055304-01 (NIH)
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Stimulant Use; Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Two groups:
  Experimental Group Control Group
Who Masked: Participant
Masking Description: All study participants are randomly assigned to a group prior to study enrollment. Participants will not be made aware of their group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Virtual Reality (Experimental): Participants in this arm will receive the following interventions:
  Virtual Reality Park Virtual Reality Avatar
  Interventions: Device: Virtual Reality
- Treatment As Usual (Placebo Comparator): Participants in this arm will receive the following interventions:
  Virtual Reality Park
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Both groups will receive a Virtual Reality Park experience, which is an empty park with no avatars. Only the experimental group will have a Virtual Reality Avatar experience, where they will see an avatar resembling themselves in a park setting.

SUMMARY:
The goal of this clinical trial is to use a novel virtual reality intervention to test for efficacy in reducing stimulant use and increasing abstinence, with concomitant increases in future self-identification, future time perspective, and delay-of-reward, in early recovering stimulant use disorder (StUD) persons. The main question[s] this trial aims to answer are:

* Will the Virtual Reality (VR) intervention decrease the number of stimulant use days?
* Will the VR intervention produce longer abstinence periods during follow-up visits?
* Will the VR intervention increase stimulant drug abstinence rates?
* Will the VR intervention increase future self-identification?
* Will the VR intervention increase self-reported future time perspective?
* Will the VR intervention increase preference for delayed rewards in a laboratory delay discounting task on the study day?
* Will the VR intervention produce gains in the behavioral effects of future self-identification, future time perspective, and delayed rewards at the 30-day and 6-month follow-ups?

Researchers will compare the experimental and control groups to see if there are differences in the results for the questions outlined above.

ELIGIBILITY:
Inclusion Criteria:

* Abstinence between ≥14 days and ≤1 year
* At least 18 years old
* Verbal endorsement of commitment to recovery
* Outpatient
* Psychotropic drugs for SUD-comorbidity
* Drug/alcohol abstinence ≥ 24 hours at the time of the study day visit
* English comprehension

Exclusion Criteria:

* Unstable medical disorders
* Less than 18 years old
* Habitual drug use
* Smell/taste disorders
* Unstable psychiatric conditions
* Extravagant/elaborate face tattoos

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduced Use of Drug Using Days | Study Day Visit; 30-day Follow-up Visit; 6-month Follow-up Visit.
  The Virtual Reality Avatar experience will reduce drug using days.
Increased Length of Abstinence | Study Day Visit; 30-day Follow-up Visit; 6-month Follow-up Visit.
  The Virtual Reality Avatar experience will increase the length of abstinence periods.
Increased (overall) Abstinence | Study Day Visit; 30-day Follow-up Visit; 6-month Follow-up Visit.
  The Virtual Reality Avatar experience will increase abstinence.
Future Self-identification | Study Day Visit; 30-day Follow-up Visit; 6-month Follow-up Visit.
  The Virtual Reality Avatar experience will increase future self-identification.
Future Time Perspective | Study Day Visit; 30-day Follow-up Visit; 6-month Follow-up Visit.
  The Virtual Reality Avatar experience will increase future time perspective.
Delayed Reward Preference | Study Day Visit; 30-day Follow-up Visit; 6-month Follow-up Visit.
  The Virtual Reality Avatar experience will increase preference for delayed rewards.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon G Oberlin, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine - Goodman Hall, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Pre-determined participant IPD will be shared in accordance with the National Institutes of Health National Data Archive requirements and upon the consent of the study participant.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be shared at the specified submission deadlines assigned by the National Institutes of Health (typically every April or October). Data will be available upon the discretion of the National Institutes of Health.
Access Criteria: No individually identifiable participant data will be submitted to the National Data Archive. All collected participant data is de-identified, and will be made available for other researchers to use upon requests submitted through the National Data Archive portal, and approval from the principal investigator.